CLINICAL TRIAL: NCT05686434
Title: Efficacy and Safety of Osimertinib Adjuvant Therapy in High-risk Stage I EGFRm NSCLC After Complete Resection(OSTAR): a Prospective, Single-arm Study
Brief Title: Osimertinib Therapy After Resection in High-risk Stage I EGFRm NSCLC (OSTAR)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-Osimertinib-001
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: NSCLC, Stage I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib adjuvant therapy group (Experimental): Patients must be enrolled within 10 weeks of complete surgical excision and receive oral Osimertinib at a dose of 80 mg once a day for a planned duration of 3 years (156 weeks).
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — This is a prospective, open, single-center, single-arm phase II clinical study with EGFR-sensitive mutations (Ex19del and L858R) identified in the central laboratory，to evaluate the efficacy and safety of adjuvant Osimertinib therapy in completely resected stage I non-squamous non-small cell lung cancer (NSCLC) with high-risk factors (solid and/or micropapillary component ≥10%, and/or airway spread).
  Other Names: Tagrisso; AZD9291

SUMMARY:
This is a prospective, open, single-center, single-arm phase II clinical study with common EGFR-sensitive mutations (Ex19del and L858R) identified in the central laboratory.To evaluate the efficacy and safety of adjuvant Osimertinib therapy in completely resected stage I non-squamous non-small cell lung cancer (NSCLC) with high-risk factors (solid and/or micropapillary component ≥10%, and/or airway spread).

DETAILED DESCRIPTION:
Patients will be tested for the status of EGFR-sensitive mutations prior to enrollment and confirmed positive by central laboratory testing.The surgically removed tumor foci will be confirmed by central laboratory pathologic examination for their pathological subtypes, solid and/or micropapillary components ≥10%, and/or STAS positive.

These patients had undergone complete resection of the tumor, and 65 patients who met the criteria for inclusion were enrolled to receive Osimertinib. Patients had to be enrolled and given Osimertinib within 10 weeks of complete resection.The dose of Osimertinib in this study was 80 mg once a day and the planned duration of treatment was 3 years (156 weeks). Patients will be evaluated for safety and efficacy at baseline, at week 12, and every 12 weeks thereafter until completion or termination of treatment. Patients were followed up every 24 weeks to 5 years (264 weeks) and annually thereafter for disease recurrence.

Overall survival (OS) was observed every 24 weeks for 5 years (264 weeks) after disease recurrence and annually thereafter.The primary endpoint of the study was 3-year DFS rate. Disease-free survival (DFS) should be calculated from the date of entry on Osimertinib to the date of disease recurrence or death.

After the primary analysis (3-year DFS rate), patients' survival status will be followed up according to the simplified study plan (OS analysis period) until the final OS analysis data is available. In the event of disease recurrence, patients will be re-staged and all sites of recurrence of NSCLC will be recorded. It will be up to the doctor to decide what treatment the patient will receive after a relapse;and cancer treatment after recurrence will be documented.Taken together, all primary, secondary, and exploratory endpoints in this study strongly describe the overall benefit of adjuvant Osimertinib in a population of patients with high-risk EGFRm+ stage I NSCLC who have been surgically completely resected.

ELIGIBILITY:
Inclusion Criteria:

1. The subject will voluntarily sign the informed consent in person, and provide the informed consent before any specific study procedures;
2. Male and female, ≥18 years old;
3. Primary non-squamous NSCLC confirmed histologically by the central laboratory;
4. Brain imaging examinations should be performed before surgery or enrollment;
5. The patient was clinically confirmed as stage I by imaging, and was staged according to the eighth edition of TNM lung cancer;
6. As confirmed by the central laboratory, the tumor contains one of the two common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), alone or in conjunction with other EGFR mutations, including T790M;
7. The primary NSCLC must be completely resected by surgery, and all lesions must be removed at the end of the surgery.All surgical margins must be negative. Lobectomy can be done with open surgery or thoracoscopic (VATS);
8. Central laboratory pathology confirmed solid and/or micropapillary component ≥10%, or STAS;
9. The interval from operation to adjuvant Osimertinib treatment is no more than 10 weeks;
10. WHO physical status score is 0~1;
11. Paraffin-embedded sections (10-15 sheets), or wax blocks or fresh frozen tissue for surgical resection of the lesion should be provided;
12. At least 2 weeks prior to initiation of the study drug, female subjects should be using highly effective contraceptive methods, pregnancy tests must be negative, and there must be no ongoing breastfeeding prior to initiation of the drug, or else one of the following criteria must be met at the time of screening to demonstrate the possibility of non-fertility:

    * Postmenopausal was defined as over 50 years of age and amenorrhea for at least 12 months after cessation of all exogenous hormone therapy.
    * Women under 50 should be considered to have stopped menstruating if they have stopped menstruating for 12 months or more after stopping exogenous hormone therapy and their LH and FSH levels are within the agency's postmenopausal range.
13. Irreversible surgical sterilization recorded by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation;Male subjects must be willing to use barrier contraception.

Exclusion Criteria:

1. Exposure to other antitumor therapies before enrollment;
2. Patients who only received segmental resection and wedge resection;
3. History of other malignancies, other than non-melanoma skin cancer, carcinoma in situ or other solid tumors that have been effectively treated, and the treating physician has determined that there is no evidence of disease recurrence for 5 years after treatment;
4. Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding, any condition that the investigator considers to be detrimental to patient participation in the study or to adherence to the protocol, or active infections including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV). Omission requirement for screening chronic diseases;
5. Any of the following cardiac criteria:

   * QTc values obtained using screening clinic ECG machines mean resting corrected QT interval (QTc) > 470 milliseconds from 3 electrocardiogram (ECG) tests,
   * Any abnormalities in rhythm, conduction, or morphology of a clinically significant resting ECG, such as left bundle branch block, third degree heart block, and second degree heart block.
   * Any factors that increase the risk of prolonged QTc or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, sudden unexplained death under 40 years of age in a first-degree relative or any concomitant medication known to prolong the QT interval.
6. Any evidence of prior history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid treatment, or active interstitial lung disease;
7. Lack of adequate bone marrow reserve or organ function (demonstrated by any of the following laboratory values: absolute neutrophil count <1.5×10⁹/L;Platelet count <100×10⁹/L;Hemoglobin <90 g/L;Alanine aminotransferase > 2.5 ULN; Aspartate aminotransferase >2.5 times ULN;Total bilirubin > 1.5 ULN;Serum creatinine >1.5 ULN with creatinine clearance <50 mL/min [as measured or calculated by Cockcroft and Gault formulas] - creatinine clearance only needs to be confirmed when creatinine >1.5 ULN);
8. History of hypersensitivity to active or inactive excipients of Osimertinib or drugs with similar chemical structures or classes to ocitinib;
9. Uncontrolled nausea and vomiting, chronic gastrointestinal illness, inability to swallow formulated drugs, or prior major bowel resection that prevents adequate absorption of Osimertinib;
10. Any evidence of corneal injury confirmed by ophthalmic examination through slit lamp evaluation;
11. The patient is pregnant or nursing;
12. History of allergy to ocitinib active or inactive excipients or drugs similar in chemical structure or class to Osimertinib;
13. If the patient is unlikely to comply with study procedures, restrictions, and requirements, the investigator judges that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-10-14 (Estimated); Study Completion 2029-10-14 (Estimated)

PRIMARY OUTCOMES:
3-year DFS rate | From date of randomisation up to approximately 5 years
  DFS is defined as time from randomization to disease recurrence (determined by CT or MRI scan and/or pathologic disease on biopsy) or death (from any cause) by investigator assessment. 3-year DFS rate is Disease-Free Survival at 3 Years.

SECONDARY OUTCOMES:
DFS | From date of randomisation up to approximately 10 years
  DFS is defined as time from randomization to disease recurrence (determined by CT or MRI scan and/or pathologic disease on biopsy) or death (from any cause) by investigator assessment.
3-year OS rate | From date of randomization up to approximately 5 years
  Defined as the percentage of patients alive at 3 years, respectively, estimated from a Kaplan Meier plot of OS at the time of the primary analysis
5-year OS rate | From date of randomization up to approximately 5 years
  Defined as the percentage of patients alive at 5 years, respectively, estimated from a Kaplan Meier plot of OS at the time of the primary analysis
OS | From date of randomization up to approximately 10 years
  OS is defined as the time from the date of randomisation until death due to any cause.
Safety and tolerability in overall population | From date of randomisation up to approximately 10 years
  AEs graded by CTCAE version 5.0
health-related quality of life and Symptoms (HRQoL) | Measured by SF-36 Questionnaire at baseline, 12 week,and then every 24 weeks until study complete, disease recurrence or other discontinuation criteria met, up to approximately 5 years.
  Change from baseline will be calculated for each domain and summary scale at each scheduled post-baseline assessment. The SF-36 includes eight domains: Physical Functioning (PF); Role Limitations-Physical (RP), Vitality (VT), General Health Perceptions (GH), Bodily Pain (BP), Social Function (SF), Role Limitations-Emotional (RE), and Mental Health (MH) and two summary scores: The Physical Component Summary (PCS) and Mental Component Summary (MCS). Final scores for each scale range from 0-100 with higher scores indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Yue, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Richeng Jiang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China